CLINICAL TRIAL: NCT03929224
Title: The Use of Medical Grade Honey in the Prevention of Bone Anchored Hearing Aid Associated Skin Breakdown
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1325595
Record Dates: First submitted 2019-03-18; First posted 2019-04-26 (Actual); Results first posted 2022-08-30 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2022-08

CONDITIONS: Skin Infection
MeSH Terms: conditions — Cellulitis | interventions — Bacitracin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bacitracin (Active Comparator): Standard care: Bone-anchored hearing aid (BAHI) abutment incision is coated in bacitracin. A healing cap is placed over the abutment and left for a week. The healing cap is removed on postoperative day 7. Patient is instructed to apply bacitracin ointment to the area for 2 weeks.
  Interventions: Drug: Bacitracin
- Medicinal honey (Experimental): Medicinal honey: Medicinal honey will be applied to the abutment site immediately after surgery. The healing cap will be placed on the BAHI site. The healing cap is removed on postoperative day 7. Patient is instructed to apply medicinal honey daily to the area for 2 weeks.
  Interventions: Drug: Medicinal honey

INTERVENTIONS:
Drug: Medicinal honey — Treat healing surgical site with medicinal honey
  Other Names: MEDIHONEY
  Arms: Medicinal honey
Drug: Bacitracin — Treat healing surgical site with bacitracin
  Arms: Bacitracin

SUMMARY:
Postoperative medicinal grade honey in post-operative care may prevent bone anchored hearing aid associated skin breakdown better than standard care of bacitracin ointment alone in adult patients.

DETAILED DESCRIPTION:
This is a prospective study. Multiple surgeons will perform the bone anchored hearing aids (BAHI) implantation surgery. Patients will be randomized to either postoperative medicinal honey or postoperative standard care of bacitracin ointment alone using a random number generator. There will be a total of two patient groups. The type of BAHI device used, laterally and the surgical technique will be recorded.

Treatment groups:

Group 1-patients undergoing BAHI implantation who will be postoperatively treated with medicinal honey.

Group 2- patients undergoing BAHI implantation who will be postoperatively treated with bacitracin ointment as standard care.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing bone-anchored hearing aid implantation surgery.

Exclusion Criteria:

* patients who are undergoing revision bone-anchored hearing surgery, history of radiation to the implantation site.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seilesh Babu, MD, Principal Investigator — Michigan Ear Institute
Locations (1):
- Ascension Providence Hospital, Novi Campus, Novi, Michigan, United States

REFERENCES:
- [Background] Costeloe A, Vandjelovic ND, Evans MA, Saraiya SS. The use of honey in cochlear implant associated wounds in pediatric patients. Int J Pediatr Otorhinolaryngol. 2018 Aug;111:80-83. doi: 10.1016/j.ijporl.2018.05.026. Epub 2018 May 24. PMID 29958620
- [Background] Faucett EA, Reghunathan S, Jacob A. Medicinal honey as treatment for skin reactions associated with bone-anchored hearing implant surgery. Laryngoscope. 2015 Jul;125(7):1720-3. doi: 10.1002/lary.25069. Epub 2014 Dec 4. No abstract available. PMID 25476170
- [Background] Bento RF, Kiesewetter A, Ikari LS, Brito R. Bone-anchored hearing aid (BAHA): indications, functional results, and comparison with reconstructive surgery of the ear. Int Arch Otorhinolaryngol. 2012 Jul;16(3):400-5. doi: 10.7162/S1809-97772012000300017. PMID 25991965
- [Background] Colquitt JL, Jones J, Harris P, Loveman E, Bird A, Clegg AJ, Baguley DM, Proops DW, Mitchell TE, Sheehan PZ, Welch K. Bone-anchored hearing aids (BAHAs) for people who are bilaterally deaf: a systematic review and economic evaluation. Health Technol Assess. 2011 Jul;15(26):1-200, iii-iv. doi: 10.3310/hta15260. PMID 21729632
- [Background] Fontaine N, Hemar P, Schultz P, Charpiot A, Debry C. BAHA implant: implantation technique and complications. Eur Ann Otorhinolaryngol Head Neck Dis. 2014 Feb;131(1):69-74. doi: 10.1016/j.anorl.2012.10.006. Epub 2013 Jul 5. PMID 23835074
- [Background] Robson V, Dodd S, Thomas S. Standardized antibacterial honey (Medihoney) with standard therapy in wound care: randomized clinical trial. J Adv Nurs. 2009 Mar;65(3):565-75. doi: 10.1111/j.1365-2648.2008.04923.x. PMID 19222654

RESULTS

PARTICIPANT FLOW:
Groups:
- Bacitracin: Standard care: BAHI abutment incision is coated in bacitracin. A healing cap is placed over the abutment and left for a week. The healing cap is removed on postoperative day 7. Patient is instructed to apply bacitracin ointment to the area for 2 weeks.
  Bacitracin: Treat healing surgical site with bacitracin
- Medicinal Honey: Medicinal honey: Medicinal honey will be applied to the abutment site immediately after surgery in addition to the bacitracin. The healing cap will be placed on the BAHI site. The healing cap is removed on postoperative day 7. Patient is instructed to apply medicinal honey daily to the area for 2 weeks.
  Medicinal honey and bacitracin: Treat healing surgical site with medicinal honey and bacitracin
Period: Overall Study
Arm/Group | Bacitracin | Medicinal Honey
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients who qualified for BAHI for single-sided deafness, conductive or mixed hearing loss on audiometric testing.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bacitracin | Medicinal Honey | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Holgers Classification of Skin Reactions at the Surgical Site Graded 0 (no Reaction) to 4 (Worse Outcome)
Description: Postoperative wound healing was compared between two groups of patients, one group had medicinal honey applied at the BAHI abutment surgical site for the first 2 weeks postoperatively, while the other group had bacitracin applied for 2 weeks. The skin at the surgical site was photographed at each time point and the photographs randomized for evaluation. The appearance of the surgical site skin was graded based on Holgers Classification by 5 separate, blinded Otolaryngologists. Holgers Classification is graded Grade 0 to Grade 4 with Grade 4 having a worse outcome. Any skin breakdown will be graded based on the Holgers Classification: Grade 0 = no reaction; Grade 1 = reddish discoloration of the skin around the implant; Grade 2 = red and moist surface of the skin around the implant; Grade 3 = formation of granulation tissue around the implant; and Grade 4 = extensive soft-tissue reaction. Holgers score was not recorded before or the day of surgery.
Time Frame: Photographs of the surgical site were taken at 1 week, 3 months and 6 months post-op.
Population: Patients qualified for BAHI: single-sided deafness, conductive or mixed hearing loss on audiometric testing.
Measure: Mean (Standard Deviation); unit: Grade
Arm/Group | Bacitracin | Medicinal Honey
Number analyzed (Participants) | 8 | 9
Grade
  1 week | 1.06 (0.78) | 0.64 (0.57)
  3 months | 0.81 (0.94) | 0.50 (0.56)
  6 months | 1.25 (1.08) | 0.68 (0.70)

2. Secondary Outcome: Number of Participants Requiring Oral Antibiotics
Description: This was determined by whether or not the patient required oral antibiotics during the 6 month follow-up period.
Time Frame: Use of oral antibiotics during the 6 months follow-up was noted.
Measure: Count of Participants; unit: Participants
Arm/Group | Bacitracin | Medicinal Honey
Number analyzed (Participants) | 8 | 9
Participants | 4 | 0

3. Secondary Outcome: Assessment of Pain at the Abutment Site Using the 0-10 Pain Scale With 0 Being no Pain At All and 10 Being the Worst Possible Pain
Description: Patient's self-reported level of pain at the abutment site was provided based on the "0 to 10 Pain Scale" with 0 being no pain at all, and 10 being the worst possible pain. Pain prior to surgery is not routinely assessed.
Time Frame: Patients self-reported their pain levels at 1 week, 3 months and 6 months post-op.
Population: The number of participants providing self-reported pain levels varied across time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bacitracin | Medicinal Honey
Number analyzed (Participants) | 8 | 9
units on a scale
  1 week: number analyzed (Participants) | 2 | 3
  1 week | 5.00 (4.24) | 2.00 (2.65)
  3 months: number analyzed (Participants) | 3 | 4
  3 months | 7.33 (2.08) | 3.00 (2.31)
  6 months: number analyzed (Participants) | 6 | 6
  6 months | 5.83 (4.12) | 0.58 (1.02)

ADVERSE EVENTS:
Time Frame: Daily for 14 days post-op and then at the 1 month, 3 month and 6 month time points
Description: For BAHI surgery, the only adverse event monitored is allergic skin reactions. Visual examination of the surgical site was performed to make sure there were no allergic skin reactions in the medicinal honey group or in the bacitracin, control group.
Groups:
- Medicinal Honey: Medicinal Honey: Medicinal honey will be applied to the abutment site immediately after surgery in addition to the bacitracin. The healing cap will be placed on the BAHI site. The healing cap is removed on postoperative day 7. Patient is instructed to apply medicinal honey daily to the area for 2 weeks.
  Medicinal honey: Treat healing surgical site with medicinal honey
Arm/Group | Bacitracin | Medicinal Honey
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9

LIMITATIONS AND CAVEATS:
The sample size was small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/24/NCT03929224/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/24/NCT03929224/ICF_001.pdf